CLINICAL TRIAL: NCT01247428
Title: A First-In-Human Trial of a New Novel DES (MiStent System) With Sirolimus and a Bioabsorbable Polymer for the Treatment of Patients With De Novo Lesions in the Native Coronary Arteries
Brief Title: First-In-Human Trial of the MiStent Drug-Eluting Stent (DES) in Coronary Artery Disease
Acronym: DESSOLVE-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Micell Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIS-FIH-2010-01
Record Dates: First submitted 2010-11-18; First posted 2010-11-24 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Drug-eluting Stent; Sirolimus
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MiStent SES (Experimental): The MiStent SES is a device/drug combination comprised of two components; a stent and a drug product (sirolimus within an absorbable polymer coating).
  Interventions: Device: MiStent SES

INTERVENTIONS:
Device: MiStent SES — The MiStent SES is a device/drug combination comprised of two components; a stent and a drug product (sirolimus within an absorbable polymer coating).

SUMMARY:
The DESSOLVE I clinical trial is to assess the safety and performance of the sirolimus-eluting MiStent SES.

DETAILED DESCRIPTION:
The DESSOLVE I clinical trial is to assess the safety and performance of the sirolimus-eluting MiStent for the treatment for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to discrete de novo lesions < 20 mm in length in the native coronary arteries with reference vessel diameters between 2.5 mm and 3.5 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients 18-85 years;
2. Stable or unstable angina pectoris, ischemia, or silent ischemia;
3. Planned single, de novo, types A, B1 and B2 coronary lesions;
4. Target lesion located in a native coronary artery;
5. Target lesion vessel diameter 2.5 to 3.5 mm amenable to treatment with a maximum 23 mm long stent;
6. Target lesion >50% diameter stenosis;
7. Patients eligible for percutaneous coronary intervention (PCI);
8. Acceptable candidate for myocardial revascularization surgery;
9. A patient may have one additional critical non-target lesion.
10. The patient will provide written informed consent.

Exclusion Criteria:

1. Female of childbearing potential not on some form of birth control with a confirmed negative pregnancy test at baseline;
2. Recent Q-wave myocardial infarction occurred <72 hours prior to the index procedure. Recent myocardial infarction with elevated levels of cardiac markers;
3. Left ventricular ejection fraction <30%;
4. Patients in cardiogenic shock;
5. Cerebrovascular accident or transient ischemic attack within 6 months;
6. Active GI bleed within three months;
7. Any prior true anaphylactic reaction to contrast agents;
8. Patient receiving/scheduled to receive chemotherapy within 30-days before or after the index procedure;
9. Patient is receiving immunosuppressive therapy or has known life-limiting immunosuppressive/autoimmune disease;
10. Renal dysfunction (creatinine > 2.0 mg/dL or 177 µmol/L);
11. Platelet count <100,000 cells/mm³ or >700,000 cells/mm³;
12. White blood cell count <3,000 cells/mm3;
13. Hepatic disease;
14. Heart transplant recipient;
15. Known contraindication to dual antiplatelet therapy;
16. Known hypersensitivity to sirolimus, cobalt-chromium, or to medications such as aspirin, heparin, and all three of the following: clopidogrel bisulfate (Plavix), ticlopidine (Ticlid), and Prasugrel (Effient);
17. Life expectancy <12 months;
18. Any major medical condition that may interfere with the optimal participation of the patient in this study;
19. Patient is currently participating/planning to participate in an investigational drug or another device study prior to completing 12-months follow-up;
20. Target vessel(s) has been treated within 10 mm proximal or distal to target lesion with any type of PCI within a year prior to index procedure;
21. Planned or actual target vessel(s) treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter prior to stent placement;
22. Previous coronary intravascular brachytherapy;
23. Planned coronary angioplasty or coronary artery bypass grafting (CABG)in the first 9 months after the index procedure;
24. Prior PCI of a non-target vessel must be at least 30 days prior to study enrollment;
25. The intent to direct stent the target lesion;
26. Angiographic Exclusion Criteria: Assessed prior to stent placement;

    * In-stent restenotic target lesion;
    * More than one lesion requiring treatment in the target vessel;
    * Target vessel diameter <2.5 mm or >3.5 mm;
    * Target lesion not amenable to treatment with a 23 mm long stent;
    * Unprotected coronary artery branch lesion (≥50% DS);
    * Target lesion located in a surgical bypass graft;
    * Total vessel occlusion;
    * Target lesion with ostial location;
    * Target lesion located in a lateral branch bifurcation >2.5mm or requiring lateral branch stenting;
    * Calcified target lesion that anticipates unsuccessful/impracticable predilation;
    * Target vessel excessive tortuosity or proximal angulation (>90 degrees);
    * Thrombus present in target vessel;
    * More than one non-target critical lesion;

Non-target lesion to be treated during the index procedure meets any of the following criteria:

* Within the target vessel;
* Within a bypass graft;
* Left main location;
* Chronic total occlusion;
* Involves a complex bifurcation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Wijns, MD, Principal Investigator — Cardiovascular Center, Onze-Lieve-Vrouwziekenhuis Aalst (OLV Hospital); John Ormiston, MD, Principal Investigator — Mercy Angiography Unit
Locations (5):
- St. Vincent's Hospital Melbourne, Melbourne, Australia
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis Aalst (OLV Hospital), Aalst
  - Ziekenhuis Oost-Limburg, Genk
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Mercy Angiography Unit - Mercy Hospital, Aukland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ormiston J, Webster M, Stewart J, Vrolix M, Whitbourn R, Donohoe D, Knape C, Lansky A, Attizzani GF, Fitzgerald P, Kandzari DE, Wijns W. First-in-human evaluation of a bioabsorbable polymer-coated sirolimus-eluting stent: imaging and clinical results of the DESSOLVE I Trial (DES with sirolimus and a bioabsorbable polymer for the treatment of patients with de novo lesion in the native coronary arteries). JACC Cardiovasc Interv. 2013 Oct;6(10):1026-34. doi: 10.1016/j.jcin.2013.05.013. Epub 2013 Sep 18. PMID 24055443
- [Result] Attizzani GF, Bezerra HG, Ormiston J, Wang W, Donohoe D, Wijns W, Costa MA. Serial assessment by optical coherence tomography of early and late vascular responses after implantation of an absorbable-coating Sirolimus-Eluting stent (from the first-in-human DESSOLVE I trial). Am J Cardiol. 2013 Nov 15;112(10):1557-64. doi: 10.1016/j.amjcard.2013.07.013. Epub 2013 Aug 29. PMID 23992957

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MiStent SES
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with symptomatic ischemic heart disease due to discrete de novo lesions < 20 mm in length in the native coronary arteries with reference vessel diameters between 2.5 mm and 3.5 mm.
Groups:
- MiStent SES: The MiStent is a device/drug combination comprised of two components; a stent and a drug product (sirolimus within an absorbable polymer coating).
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.95)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants]
  Belgium | 12
  Australia | 1
  New Zealand | 17

OUTCOME MEASURES:

1. Primary Outcome: Angiographic In-Stent Late Lumen Loss
Description: In-stent late lumen loss as measured by the angiographic core laboratory as the difference between the post-procedure minimal lumen diameters (MLD) in the treated segment (stented region) minus the MLD in the same region at follow-up.
Time Frame: 8 months
Population: Last observation used, such that patients (n=10) in the 8 month analysis is reported.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MiStent SES
Number analyzed (Participants) | 10
mm | 0.09 (0.10)

2. Secondary Outcome: Percentage of Participants Experiencing Major Adverse Cardiac Events (MACE)
Description: Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q-wave and non-Q-wave) and target vessel revascularization (TVR)
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 3.3 [0.1 to 17.2]

3. Secondary Outcome: Device Success
Description: Achievement of a final in-stent residual diameter stenosis of <50% (by QCA), using the assigned device only
Time Frame: 8 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 96.67 [82.78 to 99.92]

4. Secondary Outcome: Lesion Success
Description: Achievement of a final in-stent residual diameter stenosis of <50% (by QCA) using any percutaneous method
Time Frame: 8 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 100 [88.43 to 100]

5. Secondary Outcome: Procedural Success
Description: Achievement of a final in-stent residual diameter stenosis of <50% (by QCA) using the assigned device (including any adjunctive devices) without cardiac death, Myocardial infarction (MI) or repeat revascularization of the target lesion pre-hospital discharge
Time Frame: 8 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 100 [88.43 to 100]

6. Secondary Outcome: Total Mortality
Description: Total mortality (cardiac and non-cardiac)
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 11.6]

7. Secondary Outcome: Total Myocardial Infarction (MI)
Description: 1. Q-wave MI (QWMI): requires one of the following criteria: the development of new abnormal Q waves in ≥2 contiguous ECG leads not present on the patient's baseline (i.e., before intervention) in association with a >2x upper limit normal elevation of creatine kinase (CK) levels. In the absence of ECG data, the clinical events committee may adjudicate a Q-wave MI based on the clinical scenario and appropriate cardiac enzyme data; chest pain or other acute symptoms consistent with myocardial ischemia and new pathological Q waves in ≥2 contiguous ECG leads in the absence of timely cardiac enzyme data.
  2. Non-Q-wave MI (NQWMI): the elevation of CK levels (≥2 times ULN) with elevated CK-MB enzyme levels in the absence of new pathologic Q waves.
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 3.3 [0.1 to 17.2]

8. Secondary Outcome: Clinically-driven Target Lesion Revascularization (TLR) Rates
Description: A revascularization is considered clinically driven if angiography at follow-up shows a percent diameter stenosis ≥ 50% (Angiographic Core Laboratory QCA assessment) and if one of the following occurs:
  1. A positive history of recurrent angina pectoris, presumably related to the target vessel;
  2. Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  3. Abnormal results of any invasive functional diagnostic test (e.g., Doppler flow velocity reserve, fractional flow reserve);
  4. A target lesion revascularization (TLR) with a diameter stenosis ≥ 70% even in the absence of the above-mentioned ischemic signs or symptoms.
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 11.6]

9. Secondary Outcome: Clinically-driven Target Vessel Revascularization (TVR) Rates
Description: A revascularization is considered clinically driven if angiography at follow-up shows a percent diameter stenosis ≥ 50% (Angiographic Core Laboratory QCA assessment) and if one of the following occurs:
  1. A positive history of recurrent angina pectoris, presumably related to the target vessel;
  2. Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  3. Abnormal results of any invasive functional diagnostic test (e.g., Doppler flow velocity reserve, fractional flow reserve);
  4. A target vessel revascularization (TVR) with a diameter stenosis ≥ 70% even in the absence of the above-mentioned ischemic signs or symptoms.
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 11.6]

10. Secondary Outcome: Target Vessel Failure (TVF)
Description: Target vessel failure (TVF) is defined as the composite endpoint of:
  * cardiac death,
  * target-vessel myocardial infarction (Q wave or non-Q wave), and
  * clinically indicated target vessel revascularization
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 11.6]

11. Secondary Outcome: Target Lesion Failure (TLF)
Description: Target lesion failure (TLF) is defined as the composite endpoint of:
  * cardiac death,
  * target-lesion myocardial infarction (Q wave or non-Q wave), and
  * clinically indicated target lesion revascularization
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 11.6]

12. Secondary Outcome: Stent Thrombosis
Description: The presence of an intracoronary thrombus that originates in the stent or in the segments 5 mm proximal or distal to the stent post-procedure
Time Frame: 240 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 11.6]

13. Secondary Outcome: Angiographic Evaluation: In-stent Binary Restenosis
Description: Binary Restenosis is defined as ≥50% luminal narrowing at follow-up angiography.
Time Frame: 4 months, 6 months, 8 months
Population: Patients evaluated at 4(n=10), 6(n=10) and 8(n=10) months.
Measure: Number; unit: participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 30
participants | 0 [0 to 30.8]

14. Secondary Outcome: Angiographic Evaluation: In-stent Binary Restenosis
Description: Binary Restenosis is defined as ≥50% luminal narrowing at follow-up angiography.
Time Frame: 18 months
Population: Population includes participants from whom data was collected.
Measure: Number; unit: participants
Arm/Group | MiStent SES
Number analyzed (Participants) | 27
participants | 0 [lower limit 0.0]

15. Secondary Outcome: Intravascular Ultrasound (IVUS) Evaluation: % Neointimal Volume Obstruction
Description: % neointimal volume obstruction is defined as the neointimal volume divided by stent volume.
Time Frame: 8 months
Population: Patients evaluated at 4(n=10), 6(n=10) and 8(n=10) months. Only 25/30 patients had evaluable IVUS data.
Measure: Mean (Standard Deviation); unit: percentage of volume obstruction
Arm/Group | MiStent SES
Number analyzed (Participants) | 25
percentage of volume obstruction | 8.0 (4.4)

16. Secondary Outcome: IVUS Evaluation: % Neointimal Volume Obstruction
Description: % neointimal volume obstruction is defined as the neointimal volume divided by stent volume.
Time Frame: 18 months
Population: 20 out of 30 participants analyzed
Measure: Mean (Standard Deviation); unit: percentage of volume obstruction
Arm/Group | MiStent SES
Number analyzed (Participants) | 20
percentage of volume obstruction | 11.2 (8.1)

17. Secondary Outcome: Optical Coherence Tomography (OCT) Evaluation: % Stent Strut Uncovered
Description: % stent strut uncovered is defined as the ratio of uncovered struts to total struts in all cross-sections.
Time Frame: 8 months
Population: Patients evaluated at 4(n=10), 6(n=10) and 8(n=10) months. Only 9/30 patients had evaluable OCT at the 8 month timeframe.
Measure: Median (Full Range); unit: percentage of struts uncovered
Arm/Group | MiStent SES
Number analyzed (Participants) | 9
percentage of struts uncovered | 3.8 (2.87) [0 to 8.5]

18. Secondary Outcome: OCT Evaluation: % Stent Strut Uncovered
Description: % stent strut uncovered is defined as the ratio of uncovered struts to total struts in all cross-sections.
Time Frame: 18 M
Population: 27 out of 30 patients analyzed
Measure: Median (Full Range); unit: percentage of struts uncovered
Arm/Group | MiStent SES
Number analyzed (Participants) | 27
percentage of struts uncovered | 0 [0 to 3.4]

ADVERSE EVENTS:
Description: Regular investigator assessment.
Arm/Group | MiStent SES
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MiStent SES (N=30)
Angina pectoris (Cardiac disorders) | 2
Arteriospasm coronary (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MiStent SES (N=30)
Angina pectoris (Cardiac disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Increase tendency to bruise (Skin and subcutaneous tissue disorders) | 2
Hypertension (Surgical and medical procedures) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less